CLINICAL TRIAL: NCT00248079
Title: The Clinical Response Evaluation of the Medtronic Endeavor CR ABT-578 Eluting Coronary Stent System in De Novo Native Coronary Artery Lesions
Brief Title: The Medtronic RESOLUTE Clinical Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP069
Record Dates: First submitted 2005-11-01; First posted 2005-11-03 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Disease
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Coronary Artery Stenting — Initial implant of drug eluting stent (zotarolimus)

SUMMARY:
To evaluate the clinical safety, efficacy, and pharmacokinetics (PK) of the Endeavor Resolute Zotorolimus Eluting Coronary Stent System for the treatment of single de novo lesions in native coronary arteries with a reference vessel diameter (RVD) between 2.5 and 3.5 mm in diameter.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 18 years old
2. Patient is an acceptable candidate for percutaneous coronary intervention and emergent coronary artery bypass graft surgery
3. Patient has clinical evidence of ischemic heart disease or a positive functional study
4. Female patients of childbearing potential must have a negative pregnancy test within 7 days before the trial procedure
5. Patient or patient's legal representative has been informed of the nature of the trial and agrees to its provisions and has provided written informed consent as approved by Human Research Ethics Committee of the respective investigational site
6. Patient agrees to comply with specified follow-up evaluations and to return to the same investigational site where the procedure was performed. Patients participating in the PK sub-study must agree to the additional follow-up procedures as required by the sub-study

Exclusion Criteria:

1. Known hypersensitivity or contraindication to aspirin, heparin or bivalirudin, clopidogrel or ticlopidine, cobalt, nickel, chromium, molybdenum, polymer coating components or a sensitivity to contrast media, which cannot be adequately pre-medicated
2. History of an allergic reaction or significant sensitivity to drugs such as ABT-578, rapamycin, tacrolimus, everolimus, or any other analogue or derivative
3. Platelet count < 100,000 cells/mm³ or > 700,000 cells/mm³, or a white blood cell (WBC) count < 3,000 cells/mm³
4. Serum creatinine level > 170 micromol/L within 7 days prior to index procedure
5. Evidence of an acute myocardial infarction within 72 hours of the intended trial procedure (defined as: Q wave myocardial infarction or non-Q wave myocardial infarction having CK enzymes > 2X the laboratory upper limit of normal with the presence of an elevated CK-MB (any amount above the laboratory upper limit of normal))
6. Previous stenting anywhere in the target vessel
7. PCI of the target vessel within 30 days prior to the procedure
8. Implantation of a drug eluting stent in any non-target vessel within 30 days prior to the procedure. Implantation of a Cypher stent in any non-target vessel within 90 days prior to the procedure
9. PCI of a non-target vessel with a bare metal stent within 30 days prior to the procedure that results in any MACE event. If the bare metal stent is implanted within 72 hours prior to the procedure, a post procedural serial CK or CK-MB measurement above the investigational site's upper limit of normal (two below upper normal required for enrollment)
10. PCI of a non-target vessel within 24 hours prior to the procedure
11. Planned PCI of any vessel within 30 days post-procedure. Planned stenting of any vessel with a Cypher or Endeavor stent within 60 days post-procedure
12. Planned PCI of the target vessel within 9 months post-procedure
13. During the index procedure, the target lesion requires treatment with a device other than PTCA prior to stent placement
14. History of a stroke or transient ischemic attack within the prior 6 months
15. Active peptic ulcer or upper gastrointestinal bleeding within the prior 6 months
16. History of bleeding diathesis or coagulopathy or will refuse blood transfusions
17. Concurrent medical condition with a life expectancy of less than 12 months
18. Any previous or planned treatment of the target vessel with anti-restenotic therapies including, but not limited to brachytherapy
19. Currently participating in an investigational drug or another device trial that has not completed the primary endpoint or that clinically interferes with the current trial endpoints; or requires coronary angiography, IVUS or other coronary artery imaging procedures
20. Documented left ventricular ejection fraction < 30% at the most recent evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2005-11; Primary Completion 2007-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Late lumen loss (in-stent) as measured by quantitative coronary angiography (QCA) | 9 months

SECONDARY OUTCOMES:
Major adverse cardiac event (MACE) rate | 30 days, 4, 6, 9 & 12 months
Acute success (device, lesion, and procedure) | 4 or 9 Months
Target vessel failure (TVF) | 9 months
Target lesion revascularization (TLR) | 9 months
Neointimal hyperplastic volume and percent volume obstruction (%VO) as measured by intravascular ultrasound (IVUS) | 4 or 9 months
Pharmacokinetic parameters | last measurement at 60 days
Angiographic parameters (in-stent and in-segment) | 4 or 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Ian Meredith, Professor, Principal Investigator — Monash Medical Centre
Locations (1):
- Monash Medical Centre, Melbourne, Australia

REFERENCES:
- [Derived] Silber S, Serruys PW, Leon MB, Meredith IT, Windecker S, Neumann FJ, Belardi J, Widimsky P, Massaro J, Novack V, Yeung AC, Saito S, Mauri L. Clinical outcome of patients with and without diabetes mellitus after percutaneous coronary intervention with the resolute zotarolimus-eluting stent: 2-year results from the prospectively pooled analysis of the international global RESOLUTE program. JACC Cardiovasc Interv. 2013 Apr;6(4):357-68. doi: 10.1016/j.jcin.2012.11.006. Epub 2013 Mar 20. PMID 23523454
- [Derived] Farooq V, Vranckx P, Mauri L, Cutlip DE, Belardi J, Silber S, Widimsky P, Leon M, Windecker S, Meredith I, Negoita M, van Leeuwen F, Neumann FJ, Yeung AC, Garcia-Garcia HM, Serruys PW. Impact of overlapping newer generation drug-eluting stents on clinical and angiographic outcomes: pooled analysis of five trials from the international Global RESOLUTE Program. Heart. 2013 May;99(9):626-33. doi: 10.1136/heartjnl-2012-303368. Epub 2013 Mar 6. PMID 23468513
- [Derived] Waseda K, Ako J, Yamasaki M, Koizumi T, Sakurai R, Hongo Y, Koo BK, Ormiston J, Worthley SG, Whitbourn RJ, Walters DL, Meredith IT, Fitzgerald PJ, Honda Y. Impact of polymer formulations on neointimal proliferation after zotarolimus-eluting stent with different polymers: insights from the RESOLUTE trial. Circ Cardiovasc Interv. 2011 Jun;4(3):248-55. doi: 10.1161/CIRCINTERVENTIONS.110.957548. Epub 2011 May 17. PMID 21586691
- [Derived] Waseda K, Ako J, Yamasaki M, Koizumi T, Ormiston J, Worthley SG, Whitbourn RJ, Walters DL, Honda Y, Meredith IT, Fitzgerald PJ; RESOLUTE Trial Investigators. Short- and mid-term intravascular ultrasound analysis of the new zotarolimus-eluting stent with durable polymer - results from the RESOLUTE trial -. Circ J. 2010 Oct;74(10):2097-102. doi: 10.1253/circj.cj-10-0063. Epub 2010 Aug 3. PMID 20689221
- [Derived] Remak E, Manson S, Hutton J, Brasseur P, Olivier E, Gershlick A. Cost-effectiveness of the Endeavor stent in de novo native coronary artery lesions updated with contemporary data. EuroIntervention. 2010 Feb;5(7):826-32. doi: 10.4244/eijv5i7a138. PMID 20142198
- [Derived] Meredith IT, Worthley S, Whitbourn R, Walters DL, McClean D, Horrigan M, Popma JJ, Cutlip DE, DePaoli A, Negoita M, Fitzgerald PJ; RESOLUTE Investigators. Clinical and angiographic results with the next-generation resolute stent system: a prospective, multicenter, first-in-human trial. JACC Cardiovasc Interv. 2009 Oct;2(10):977-85. doi: 10.1016/j.jcin.2009.07.007. PMID 19850258